CLINICAL TRIAL: NCT03475225
Title: Effect of the Treatment of Vitamin D Deficiency in Drug-resistant Epilepsy
Brief Title: Vitamine D in Drug Resistant Epilepsy
Acronym: EPI-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: APHP (Other); FFRE (Unknown); LFCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D16-P15
Record Dates: First submitted 2017-12-26; First posted 2018-03-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Drug Resistant Epilepsy
Keywords: Epilepsy; Drug-resistance; Vitamin D deficiency; Metabolism; Controlled study antiepileptic drugs
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Double blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Drug resistant epilepsy patients with proved Vitamin D deficiency (Serum vitamin D level <30ng/ml) Cholecalciferol. 5 doses of cholecalciferol (100 000 IU) in 3 months than 1 dose of cholecalciferol (100 000 IU) per month during 6 months
  Interventions: Drug: Cholecalciferol
- Control Arm (Placebo Comparator): Drug resistant epilepsy patients with proved Vitamin D deficiency (Serum vitamin D level<30ng/ml) Placebo than cholecalciferol. 5 doses of placebo in 3 months than 5 doses of cholecalciferol (100 000 IU) in 3 months than 1 dose of cholecalciferol (100 000 IU) per month during 3 months.
  Interventions: Drug: Placebo Oral

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol delivery
  Arms: Experimental Arm
Drug: Placebo Oral — manufactured to mimic Cholecalciferol
  Arms: Control Arm

SUMMARY:
Almost all patients with epilepsy living in the region of Paris have vitamin D deficiency, which is severe in 1/3 of the cases. The impact of this deficiency on epilepsy is unknown, despite the suggested benefits of vitamin D therapy including better seizure control and improvement of comorbidities (fatigue, anxiety, depression) in drug-resistant patients. Recommendations for vitamin D supplementation based on the serum level in the general population cannot be applied to patients with epilepsy due to interference of antiepileptic drugs in the vitamin D metabolism. Animal models, mechanisms of action studies and ecological information provide objective data for a direct antiepileptic effect of vitamin D. Human studies seem to confirm the antiepileptic effect of vitamin D but there are no controlled studies on large populations. The investigators aim to assess prospectively the effect of the treatment of vitamin D deficiency providing a high level of evidence. The investigators propose a multicentre placebo controlled randomized double-blind study, testing vitamin D supplementation against placebo in 400 drug-resistant patients to assess the short-term (3 months) and long-term (1 year) benefits on epilepsy. The investigators hypothesize that the treatment of vitamin D deficiency will result in significant reduction of seizure frequency, and improvement of comorbid symptoms as well as quality of life. The impact on the care of patients is important because better epilepsy control allows reduction of the antiepileptic drugs and side effects. This again is a key for the recovery of social and professional activities, and reduction of costs related to the disease.

DETAILED DESCRIPTION:
The goal of this study is to establish the effect of the compensation of vitamin D deficiency in the treatment of drug-resistant epilepsy with a high level of evidence in a large population. For that, the investigator aim to perform a controlled multicentre prospective double-blind randomized study in 400 patients.

Experimental design

After a reference period for the collection of clinical data and seizure frequency, all eligible patients will undergo biological analyses including serum vitamin D levels, calcium, creatinine and albumin. In case of proven deficiency (25(OH)D <30ng/mL), patients will be randomized into two arms:

Experimental group: drug-resistant epileptic patients supplemented with vitamin D. The vitamin D administered corresponds to the scheme described below. Control group: drug-resistant epileptic patients supplemented with placebo, administered placebo dose is equal to therapeutic dosing scheme of vitamin D. Randomization will be centralized and stratified by center (considering local disparities) and according to the results of serum level, retaining the threshold of 10ng/mL to define severe deficiency, 20 ng/mL for moderate deficiency and 30 ng/mL for slight deficiency of vitamin D.

The drug evaluated is vitamin D3 (cholecalciferol), administered in the form of oral solution (2 mL) containing 100,000 IU, manufactured by the laboratory CRINEX and marketed under the name UVEDOSE®. The therapeutic indication is the treatment and/or prophylaxis of vitamin D deficiency. The usual supplementation in adult is 1 to 2 doses per month depending on the severity of the deficiency, the maintenance ranging from 1 dose every month or every 2 to 3 months.

Administration in the experimental group and control group The supplementation scheme is based on the usual recommendations but does not take into account the severity of the initial deficiency, that would be impossible to implement in the context of a double-blind study (with in particular the need to adapt each placebo dose in the control group, risking the feasibility study). To address this potential bias, the investigators choice a supplementation scheme corresponding to a moderate deficiency (25(OH)D >10 and <20ng/mL) considering that this is the most common in clinical practice and there is no risk of overdose for 25(OH)D level between 20 and 30ng/mL.

The dosing schedule is as follows:

UVEDOSE: 1 dose of 100,000 IU every 15 days for 2 months, then 100,000 IU the 3rd month (5 doses during the first 3 months). Dosage of 25(OH)D will be conducted at 3 and 6 months in order to verify the compensation of the initial deficiency and to avoid the risk of overdose. Monitoring of serum calcium, albumin and creatinine will be performed at the same time. Maintenance therapy in the treatment group will be set at 100,000 IU per month for 6 months (11 doses for 12 months followup). After the blind period, the same will be applied to the control group (5 doses in 3 months and 1 dose per month for 3 months, 8 doses for 12 months follow-up).

Apart from an overdose, no side effects are expected. An overdose of vitamin D may be suspected in case of occurrence of one or more of the following signs: headache, asthenia, anorexia, weight loss; nausea, vomiting; polyuria, polydipsia, dehydration; high blood pressure; calcium lithiasis; renal insufficiency. Biological signs reflecting the vitamin D overdose are hypercalcemia with hypercalciuria. Serum levels of 25(OH)D from 100 to 150 ng/mL are exceptionally accompanied by hypercalcemia. High risk of hypercalcemia with clinical consequences are reported for levels around 250ng/mL whereas no toxic effects are described for serum levels <150 ng/mL. To avoid any risk, the supplementation will be stopped if the dosage of 25(OH)D is >100ng/mL and/or serum calcium levels >2.70mmol/l; if the serum calcium is >2.60 and <2.70mmol/l, a control will be done and the treatment stopped if >2.60mmol/L. Vitamine D treatment will be stopped also if creatinine is >200μmol/L. Vitamin D causes no known drug interactions. However its metabolism is accelerated when combined with enzyme-inducing drugs, including antiepileptic drugs.

The entire treatment will be provided to each patient using a kit of 5 doses of UVEDOSE after randomization in the experimental group and the unblinding in the control group according to the protocol established. The treatment scheme will be clearly explained and dates of treatment indicated on the attached schedule. Maintenance therapy will be provided on the same terms.

Patients will note on this calendar the effective date of each dose and bring empty containers during the visit at 3 months, 6 months and 12 months. The labeling will be performed by the laboratory CRINEX, the kits will be delivered to pharmacy centers. The pharmacy of each participating center will handle the management of returns and the destruction of processing units. Patients in the control group will receive placebo of vitamin D in the same manner as experimental patients.

The study entails a screening-visit followed by a 3 months reference period, an inclusion visit followed by randomization, two follow-up visits (3 and 6 months) and an end-study visit at 12 months. The duration of study for each patient is 12 months following the 3 months reference-phase. The double-blind phase is between the randomization (V1) and the 3 month visit (V2), followed by a 9 month open phase for the 2 groups Eventually, all patients with a vitamin D deficiency will be compensated with a 3-month higher dose treatment phase and a 6-month maintenance phase for the experimental group. The control group will receive the placebo for 3 months, then a vitamin D treatment including a 3-month higher dose and a 3 month maintenance phase.

The duration of the inclusions is scheduled for 12 months, for research duration of 24 months. All eligible patients who meet ILAE (International League Against Epilepsy) criteria of drug-resistance and inclusion criteria will be informed of the opportunity to participate in this research. If accepted, the participants will be asked to fill out a precise seizure diary for 3 months before their inclusion in the study (V0). The antiepileptic treatment should not be changed during the reference period. The patient cannot receive vitamin D during this period.

Inclusion visit (V1):

After obtaining informed consent and verification of inclusion criteria, seizure frequency is noted and determination of serum 25(OH)D level is done. The vitamin D serum concentration is determined with the same technic in each center (immunoluminometric CLIA (Chemiluminescence Immunoassay Analyzer) - Liaison XL). The concentration serum calcium, albumin and creatinine is determined at the biochemistry laboratory of the participating center. The self-questionnaires (Fatigue impact scale : FIS, Hospital anxiety depression scale :HAD, Quality of life in epilepsy : QOLIE 31) are completed and handed to the investigator. Clinical and demographic data are collected on the case report. After receipt of 25(OH)D level results, patients in whom deficiency is objectified (25(OH)D <30ng/mL) are randomized between control and experimental group. It is expected 10% of non-deficient patients who are not randomized and followed out of the protocol. Treatment appropriate to the protocol for each group (vitamin D or placebo) is delivered by the center pharmacy. The results of biology (serum calcium, albumin, creatinine) are first referred to the investigator, the treatment being delivered in absence of contra-indication (see above).

3 month-visit (V2): Clinical examination, seizure frequency, determination of 25(OH)D levels, serum calcium, albumin, creatinine) and scales (FIS, HAD, QOLIE 31); monitoring of compliance (ratio of packaging and check-up of dates); lifting of the blinding phase. Introduction of vitamin D supplementation in the placebo group according to the initial plan, pursuit of vitamin D supplementation in the experimental group, stop if the serum level is>100 ng/mL and/or serum calcium>2.70mmol/L and/or creatinine>200 μmol/L. Control of serum calcium if between 2.60 and 2.70 mmol/L, stop if> 2.60 mmol/L.

6 month-visit (V3): similar to V2, maintenance supplementation in the 2 groups: 1 dose per month for 3 months, except if biological contraindication.

End-study visit (V4, 12 months) similar to V1-V2, vitamin D trial stop. In case of deterioration of the clinical situation requiring modification of the antiepileptic treatment (excluding one-time treatment with benzodiazepines), the patient will be considered not-responder but will not be excluded from the study. The seizure frequency in this case for the primary judgment criterion will be the one before the treatment change (LOCF method).

ELIGIBILITY:
Inclusion Criteria:

* Age> 15 years
* Drug-resistant epilepsy (see definition above)
* Having at least 6 unprovoked seizures in the previous 3 months
* Epilepsy syndrome unequivocally established
* Ability to reliably quantify the seizure frequency
* Antiepileptic treatment stable for 3 months prior to inclusion
* No vitamin D treatment in the 6 months prior to inclusion vitamin D supplemental diet
* Medication compliance (confirmed by plasma levels if available)
* Agreeing to participate in the study
* Having a social insurance
* Parental agreement if patient below the age to be able to give consent (or guardian if protected adult)

Exclusion Criteria:

* Progressive brain pathology
* Status epilepticus in the 2 years prior to inclusion,
* epilepsy surgery planned in the current year
* Pregnancy or breast-feeding
* Treatments influencing the metabolism of vitamin D other than anticoagulants (rifamycin, isoniazid, ketoconazole, 5-FU fluorouracil), leucovorin)
* Known hypersensitivity to vitamin D, patients with a history of granulomatosis (especially sarcoidosis)
* Contraindication to treatment with Uvedose referring to the summary of product characteristics
* Current or past hypercalcemia or situations accompanied by increased vulnerability to hypercalcemia as arrhythmia or digitalis therapy, subjects with calcium lithiasis
* Moderate renal impairment with creatinine clearance <60 mL/mn assessed by MDRD (Modification of Diet in Renal Disease)
* Participation in other studies of other experimental drugs within 30 days before enrollment in the study
* Abuse of alcohol or drugs

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage reduction of the seizure frequency | After 3 months of treatment of vitamin D deficiency
  With respect to the reference period

SECONDARY OUTCOMES:
Effect on Fatigue scores : Modified Fatigue Impact Scale (M-FIS) | 3, 6 and 12 months
  Total score at baseline and after Vitamin D treatment (range 0-200; higher values=worse outcome)
Effect anxiety-depression : Hospital anxiety depression scale (HAD) | 3, 6 and 12 months
  Total score at baseline and after Vitamin D treatment (range 0-42; higher values=worse outcome)
Quality of Life in Epilepsy: (QOLIE 31) including 7 subscores: global score calculated on the basis on the mean of each subscore | 3, 6 and 12 months
  Global score at baseline and after Vitamin D treatment (the higher score, the better outcome)
Relationship between serum vitamin D levels and seizure frequency reduction after vitamin D treatment | 3, 6 and 12 months
  Vitamin D levels and percentage reduction in the seizure frequency compared to the reference period
Relationship between serum vitamin D levels and seizure frequency reduction after vitamin D treatment | 3, 6 and 12 months.
  Vitamin D level and type of AED (enzyme inducer versus non enzyme inducer drugs)
Relationship between serum vitamin D level and the type and dosage of antiepileptic drugs (AED) | Baseline
  Vitamin D level and dose of AED (low dose versus high dose of enzyme inducer drugs)
Responder rate | 3, 6 and 12 months.
  Responder rate after Vitamin D treatment. Percentage of patients having a reduction of at least 50% of the seizure frequency
Remission rate after Vitamin D treatment | 3, 6 and 12 months.]
  Percentage of patients without any seizure (seizure freedom)
Effect of Vitamin D according to epilepsy type | 3, 6 and 12 months
  Responder rate in focal and generalized epilepsy
Effect of Vitamin D according to epilepsy severity | 3, 6 and 12 months
  Percentage of reduction of secondary generalized seizures and epileptic falls in respect to the reference period

CONTACTS AND LOCATIONS:
Overall Officials: CHASSOUX Francine, MD, Principal Investigator — Centre Hospitalier Sainte-Anne - 1, rue Cabanis 75014 Paris FRANCE
Locations (2):
- France (2):
  - Hôpital Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Sainte Anne, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baxendale S. Seeing the light? Seizures and sunlight. Epilepsy Res. 2009 Mar;84(1):72-6. doi: 10.1016/j.eplepsyres.2008.11.015. Epub 2009 Jan 13. PMID 19144500
- [Background] Beyenburg S, Stavem K, Schmidt D. Placebo-corrected efficacy of modern antiepileptic drugs for refractory epilepsy: systematic review and meta-analysis. Epilepsia. 2010 Jan;51(1):7-26. doi: 10.1111/j.1528-1167.2009.02299.x. Epub 2009 Sep 10. PMID 19744114
- [Background] Borowicz KK, Morawska M, Furmanek-Karwowska K, Luszczki JJ, Czuczwar SJ. Cholecalciferol enhances the anticonvulsant effect of conventional antiepileptic drugs in the mouse model of maximal electroshock. Eur J Pharmacol. 2007 Nov 14;573(1-3):111-5. doi: 10.1016/j.ejphar.2007.07.002. Epub 2007 Jul 10. PMID 17643415
- [Background] Callaghan B, Schlesinger M, Rodemer W, Pollard J, Hesdorffer D, Allen Hauser W, French J. Remission and relapse in a drug-resistant epilepsy population followed prospectively. Epilepsia. 2011 Mar;52(3):619-26. doi: 10.1111/j.1528-1167.2010.02929.x. Epub 2011 Jan 26. PMID 21269287
- [Background] Carbone LD, Johnson KC, Robbins J, Larson JC, Curb JD, Watson K, Gass M, Lacroix AZ. Antiepileptic drug use, falls, fractures, and BMD in postmenopausal women: findings from the women's health initiative (WHI). J Bone Miner Res. 2010 Apr;25(4):873-81. doi: 10.1359/jbmr.091027. PMID 19839772
- [Background] Carnes J, Quinn S, Nelson M, Jones G, Winzenberg T. Intermittent high-dose vitamin D corrects vitamin D deficiency in adolescents: a pilot study. Eur J Clin Nutr. 2012 Apr;66(4):530-2. doi: 10.1038/ejcn.2011.204. Epub 2011 Dec 21. PMID 22190133
- [Background] Cavalier E, Fache W, Souberbielle JC. A Randomised, Double-Blinded, Placebo-Controlled, Parallel Study of Vitamin D3 Supplementation with Different Schemes Based on Multiples of 25,000 IU Doses. Int J Endocrinol. 2013;2013:327265. doi: 10.1155/2013/327265. Epub 2013 Jan 28. PMID 23431293
- [Background] Christensen J, Vestergaard M, Mortensen PB, Sidenius P, Agerbo E. Epilepsy and risk of suicide: a population-based case-control study. Lancet Neurol. 2007 Aug;6(8):693-8. doi: 10.1016/S1474-4422(07)70175-8. PMID 17611160
- [Background] Christiansen C, Rodbro P, Sjo O. "Anticonvulsant action" of vitamin D in epileptic patients? A controlled pilot study. Br Med J. 1974 May 4;2(5913):258-9. doi: 10.1136/bmj.2.5913.258. PMID 4207965
- [Background] Devaux B, Chassoux F, Guenot M, Haegelen C, Bartolomei F, Rougier A, Bourgeois M, Colnat-Coulbois S, Bulteau C, Sol JC, Kherli P, Geffredo S, Reyns N, Vinchon M, Proust F, Masnou P, Dupont S, Chabardes S, Coubes P. [Epilepsy surgery in France]. Neurochirurgie. 2008 May;54(3):453-65. doi: 10.1016/j.neuchi.2008.02.041. Epub 2008 May 7. French. PMID 18466930
- [Background] Duhamel JF, Zeghoud F, Sempe M, Boudailliez B, Odievre M, Laurans M, Garabedian M, Mallet E. [Prevention of vitamin D deficiency in adolescents and pre-adolescents. An interventional multicenter study on the biological effect of repeated doses of 100,000 IU of vitamin D3]. Arch Pediatr. 2000 Feb;7(2):148-53. doi: 10.1016/s0929-693x(00)88084-7. French. PMID 10701059
- [Background] Duncan JS, Sander JW, Sisodiya SM, Walker MC. Adult epilepsy. Lancet. 2006 Apr 1;367(9516):1087-1100. doi: 10.1016/S0140-6736(06)68477-8. PMID 16581409
- [Background] Eyles DW, Smith S, Kinobe R, Hewison M, McGrath JJ. Distribution of the vitamin D receptor and 1 alpha-hydroxylase in human brain. J Chem Neuroanat. 2005 Jan;29(1):21-30. doi: 10.1016/j.jchemneu.2004.08.006. PMID 15589699
- [Background] Fazel S, Wolf A, Langstrom N, Newton CR, Lichtenstein P. Premature mortality in epilepsy and the role of psychiatric comorbidity: a total population study. Lancet. 2013 Nov 16;382(9905):1646-54. doi: 10.1016/S0140-6736(13)60899-5. Epub 2013 Jul 22. PMID 23883699
- [Background] Fertig E, Fureman BE, Bergey GK, Brodie MA, Hesdorffer DC, Hirtz D, Kossoff EH, LaFrance WC Jr, Versavel M, French J; National Institute of Neurological Disorders and Stroke. Inclusion and exclusion criteria for epilepsy clinical trials-recommendations from the April 30, 2011 NINDS workshop. Epilepsy Res. 2014 Jul;108(5):825-32. doi: 10.1016/j.eplepsyres.2014.02.011. Epub 2014 Mar 1. PMID 24702822
- [Background] Hamelin S, Kahane P, Vercueil L. Fatigue in epilepsy: a prospective inter-ictal and post-ictal survey. Epilepsy Res. 2010 Oct;91(2-3):153-60. doi: 10.1016/j.eplepsyres.2010.07.006. Epub 2010 Aug 12. PMID 20708384
- [Background] Hermann BP, Seidenberg M, Dow C, Jones J, Rutecki P, Bhattacharya A, Bell B. Cognitive prognosis in chronic temporal lobe epilepsy. Ann Neurol. 2006 Jul;60(1):80-7. doi: 10.1002/ana.20872. PMID 16802302
- [Background] Hesdorffer DC. Motor vehicle accidents, suicides, and assaults in epilepsy: a population-based study. Neurology. 2011 Oct 25;77(17):1653; author reply 1653-4. doi: 10.1212/WNL.0b013e318230b17e. No abstract available. PMID 22025462
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Hollo A, Clemens Z, Kamondi A, Lakatos P, Szucs A. Correction of vitamin D deficiency improves seizure control in epilepsy: a pilot study. Epilepsy Behav. 2012 May;24(1):131-3. doi: 10.1016/j.yebeh.2012.03.011. Epub 2012 Apr 11. PMID 22503468
- [Background] Hollo A, Clemens Z, Lakatos P. Epilepsy and vitamin D. Int J Neurosci. 2014 Jun;124(6):387-93. doi: 10.3109/00207454.2013.847836. Epub 2013 Nov 7. PMID 24063762
- [Background] Kalueff AV, Minasyan A, Tuohimaa P. Anticonvulsant effects of 1,25-dihydroxyvitamin D in chemically induced seizures in mice. Brain Res Bull. 2005 Sep 30;67(1-2):156-60. doi: 10.1016/j.brainresbull.2005.06.022. PMID 16140175
- [Background] Kalueff AV, Minasyan A, Keisala T, Kuuslahti M, Miettinen S, Tuohimaa P. Increased severity of chemically induced seizures in mice with partially deleted Vitamin D receptor gene. Neurosci Lett. 2006 Feb 6;394(1):69-73. doi: 10.1016/j.neulet.2005.10.007. Epub 2005 Oct 25. PMID 16256271
- [Background] Kanner AM. Depression in epilepsy: prevalence, clinical semiology, pathogenic mechanisms, and treatment. Biol Psychiatry. 2003 Aug 1;54(3):388-98. doi: 10.1016/s0006-3223(03)00469-4. PMID 12893113
- [Background] Kanner AM. The treatment of depressive disorders in epilepsy: what all neurologists should know. Epilepsia. 2013 Mar;54 Suppl 1:3-12. doi: 10.1111/epi.12100. PMID 23458461
- [Background] Kanner AM. Do psychiatric comorbidities have a negative impact on the course and treatment of seizure disorders? Curr Opin Neurol. 2013 Apr;26(2):208-13. doi: 10.1097/WCO.0b013e32835ee579. PMID 23429545
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Kwan P, Schachter SC, Brodie MJ. Drug-resistant epilepsy. N Engl J Med. 2011 Sep 8;365(10):919-26. doi: 10.1056/NEJMra1004418. No abstract available. PMID 21899452
- [Background] Lazzari AA, Dussault PM, Thakore-James M, Gagnon D, Baker E, Davis SA, Houranieh AM. Prevention of bone loss and vertebral fractures in patients with chronic epilepsy--antiepileptic drug and osteoporosis prevention trial. Epilepsia. 2013 Nov;54(11):1997-2004. doi: 10.1111/epi.12351. Epub 2013 Sep 6. PMID 24010637
- [Background] Mann MW, Pons G. [Drug resistance in partial epilepsy: epidemiology, mechanisms, pharmacogenetics and therapeutical aspects]. Neurochirurgie. 2008 May;54(3):259-64. doi: 10.1016/j.neuchi.2008.02.018. Epub 2008 Apr 15. French. PMID 18417170
- [Background] Menon B, Harinarayan CV. The effect of anti epileptic drug therapy on serum 25-hydroxyvitamin D and parameters of calcium and bone metabolism--a longitudinal study. Seizure. 2010 Apr;19(3):153-8. doi: 10.1016/j.seizure.2010.01.006. Epub 2010 Feb 7. PMID 20144552
- [Background] McGrath J, Feron F, Eyles D, Mackay-Sim A. Vitamin D: the neglected neurosteroid? Trends Neurosci. 2001 Oct;24(10):570-2. doi: 10.1016/s0166-2236(00)01949-4. No abstract available. PMID 11576669
- [Background] Picot MC, Jaussent A, Neveu D, Kahane P, Crespel A, Gelisse P, Hirsch E, Derambure P, Dupont S, Landre E, Chassoux F, Valton L, Vignal JP, Marchal C, Lamy C, Semah F, Biraben A, Arzimanoglou A, Petit J, Thomas P, Macioce V, Dujols P, Ryvlin P. Cost-effectiveness analysis of epilepsy surgery in a controlled cohort of adult patients with intractable partial epilepsy: A 5-year follow-up study. Epilepsia. 2016 Oct;57(10):1669-1679. doi: 10.1111/epi.13492. Epub 2016 Sep 5. PMID 27595433
- [Background] Pierrot-Deseilligny C, Souberbielle JC. Is hypovitaminosis D one of the environmental risk factors for multiple sclerosis? Brain. 2010 Jul;133(Pt 7):1869-88. doi: 10.1093/brain/awq147. PMID 20584945
- [Background] Pierrot-Deseilligny C, Souberbielle JC. Widespread vitamin D insufficiency: A new challenge for primary prevention, with particular reference to multiple sclerosis. Presse Med. 2011 Apr;40(4 Pt 1):349-56. doi: 10.1016/j.lpm.2011.01.003. Epub 2011 Feb 17. PMID 21333483
- [Background] Procopio M, Marriott PK, Williams P. Season of birth: aetiological implications for epilepsy. Seizure. 1997 Apr;6(2):99-105. doi: 10.1016/s1059-1311(97)80062-3. PMID 9153721
- [Background] Saggese G, Vierucci F, Boot AM, Czech-Kowalska J, Weber G, Camargo CA Jr, Mallet E, Fanos M, Shaw NJ, Holick MF. Vitamin D in childhood and adolescence: an expert position statement. Eur J Pediatr. 2015 May;174(5):565-76. doi: 10.1007/s00431-015-2524-6. Epub 2015 Apr 2. PMID 25833762
- [Background] Schiller Y, Najjar Y. Quantifying the response to antiepileptic drugs: effect of past treatment history. Neurology. 2008 Jan 1;70(1):54-65. doi: 10.1212/01.wnl.0000286959.22040.6e. PMID 18166707
- [Background] Schmidt D, Schachter SC. Drug treatment of epilepsy in adults. BMJ. 2014 Feb 28;348:g254. doi: 10.1136/bmj.g254. PMID 24583319
- [Background] Semah F, Picot MC, Adam C, Broglin D, Arzimanoglou A, Bazin B, Cavalcanti D, Baulac M. Is the underlying cause of epilepsy a major prognostic factor for recurrence? Neurology. 1998 Nov;51(5):1256-62. doi: 10.1212/wnl.51.5.1256. PMID 9818842
- [Background] Siegel A, Malkowitz L, Moskovits MJ, Christakos S. Administration of 1,25-dihydroxyvitamin D3 results in the elevation of hippocampal seizure threshold levels in rats. Brain Res. 1984 Apr 23;298(1):125-9. doi: 10.1016/0006-8993(84)91153-3. PMID 6547070
- [Background] Sisodiya SM, Lin WR, Harding BN, Squier MV, Thom M. Drug resistance in epilepsy: expression of drug resistance proteins in common causes of refractory epilepsy. Brain. 2002 Jan;125(Pt 1):22-31. doi: 10.1093/brain/awf002. PMID 11834590
- [Background] Souberbielle JC, Benhamou CL, Cortet B, Rousiere M, Roux C, Abitbol V, Audran M, Bachetta J, Beauchet O, Blain H, Breuil V, Briot K, Brunet P, Chanson P, Cormier C, Courbebaisse M, Fardellone P, Fouque D, Friedlander G, Gauvain JB, Groussin L, Houillier P, Jacot W, Jean G, Kamenicky P, Lafage-Proust MH, Legrand E, Levy-Weil F, Linglart A, Mallet E, Marcelli C, Maruani G, Montagnon F, Personne V, Prie D, Raynaud-Simon A, Rolland Y, Salle B, Sault C, Schott AM, Thervet E, Urena-Torres P, Viard JP, Weryha G, Pierrot-Deseilligny C, Young J, Thomas T. [HAS report on vitamin D measurement: don't go from an extreme situation to another as extreme situation]. Presse Med. 2014 Jan;43(1):5-8. doi: 10.1016/j.lpm.2013.12.005. No abstract available. French. PMID 24439118
- [Background] Steinhoff BJ. Efficacy of perampanel: a review of pooled data. Epilepsia. 2014 Jan;55 Suppl 1:9-12. doi: 10.1111/epi.12493. PMID 24400691
- [Background] Teagarden DL, Meador KJ, Loring DW. Low vitamin D levels are common in patients with epilepsy. Epilepsy Res. 2014 Oct;108(8):1352-6. doi: 10.1016/j.eplepsyres.2014.06.008. Epub 2014 Jul 6. PMID 25060996
- [Background] Tellez-Zenteno JF, Patten SB, Jette N, Williams J, Wiebe S. Psychiatric comorbidity in epilepsy: a population-based analysis. Epilepsia. 2007 Dec;48(12):2336-44. doi: 10.1111/j.1528-1167.2007.01222.x. Epub 2007 Jul 28. PMID 17662062
- [Background] Vestergaard P, Rejnmark L, Mosekilde L. Fracture risk associated with use of antiepileptic drugs. Epilepsia. 2004 Nov;45(11):1330-7. doi: 10.1111/j.0013-9580.2004.18804.x. PMID 15509233
- [Background] Vidailhet M, Mallet E, Bocquet A, Bresson JL, Briend A, Chouraqui JP, Darmaun D, Dupont C, Frelut ML, Ghisolfi J, Girardet JP, Goulet O, Hankard R, Rieu D, Simeoni U, Turck D; Comite de nutrition de la Societe francaise de pediatrie. Vitamin D: still a topical matter in children and adolescents. A position paper by the Committee on Nutrition of the French Society of Paediatrics. Arch Pediatr. 2012 Mar;19(3):316-28. doi: 10.1016/j.arcped.2011.12.015. Epub 2012 Jan 27. PMID 22284232
- [Background] Wassenaar M, Leijten FS, Egberts TC, Moons KG, Uijl SG. Prognostic factors for medically intractable epilepsy: a systematic review. Epilepsy Res. 2013 Oct;106(3):301-10. doi: 10.1016/j.eplepsyres.2013.06.013. Epub 2013 Jul 20. PMID 23880113
- [Background] de Zelicourt M, de Toffol B, Vespignani H, Laurendeau C, Levy-Bachelot L, Murat C, Fagnani F. Management of focal epilepsy in adults treated with polytherapy in France: the direct cost of drug resistance (ESPERA study). Seizure. 2014 May;23(5):349-56. doi: 10.1016/j.seizure.2014.01.016. Epub 2014 Jan 30. PMID 24560531
- [Derived] Chassoux F, Navarro V, Quirins M, Laurent A, Gavaret M, Cousyn L, Crepon B, Landre E, Marchi A, Soufflet C, Rusu-Devaux V, Mancusi RL, Piketty ML, Souberbielle JC. Vitamin D deficiency and effect of treatment on seizure frequency and quality of life parameters in patients with drug-resistant epilepsy: A randomized clinical trial. Epilepsia. 2024 Sep;65(9):2612-2625. doi: 10.1111/epi.18050. Epub 2024 Jul 9. PMID 38980968